CLINICAL TRIAL: NCT06959511
Title: Neoadjuvant Treatment With Zanzalintinib for Advanced Thyroid Cancer
Brief Title: Zanzalintinib for the Treatment of Advanced Thyroid Cancer Before Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0308; NCI-2025-03105 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Neoadjuvant Treatment; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant with Zanzalintinib Followed by Surgery (Experimental): Zanzalintinib 100 mg orally once daily on Days 1 to 28 of a 28-day cycle.
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — Given by po

SUMMARY:
To look at the effectiveness of zanzalintinib, followed by surgery, in treating advanced thyroid cancer. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Primary Objectives

• To evaluate the efficacy of neoadjuvant zanzalintinib in DTC, non-RET-mutated MTC, and poorly differentiated thyroid cancer (PDTC) by overall objective response rate (overall ORR), defined as the proportion of participants who have a minor response (MR), partial response (PR), or complete response (CR) per RECIST. Participants with locally invasive extrathyroidal and/or extra nodal DTC, non- RET-mutated MTC or PDTC who have high surgical morbidity/complexity based on baseline radiographic assessment (as measured by Thyroid Neck Surgical Morbidity/Complexity Scoring, see Section 3.2.1), will be eligible for the study.

Hypothesis: Neoadjuvant administration of zanzalintinib will result in acceptable overall ORR (MR+PR+CR rate) for participants with locoregionally advanced DTC and non-RETmutated MTC, ultimately allowing patients to safely undergo complete gross surgical tumor resection with less surgical morbidity.

Secondary Objectives

* To evaluate the efficacy of neoadjuvant zanzalintinib in DTC, non-RET-mutated MTC or PDTC by objective response rate (ORR) per modified neck RECIST.
* To evaluate the safety profile of neoadjuvant zanzalintinib in thyroid cancer.
* To evaluate the efficacy of neoadjuvant zanzalintinib on progression-free survival (PFS), including overall PFS and locoregional PFS.
* To measure changes in expected and actual thyroid neck surgical morbidity/complexity scoring before and after zanzalintinib treatment.
* To evaluate the efficacy of neoadjuvant zanzalintinib by surgical margin status.

Exploratory Objectives

* To define and measure changes of patient-reported outcomes (PROs) and quality of life (QOL) as measured by MDASI-HN and EQ-5D in participants who receive zanzalintinib treatment.
* To evaluate the efficacy of neoadjuvant zanzalintinib by pathologic response.
* To evaluate the efficacy of neoadjuvant zanzalintinib by PET metabolic response.

ELIGIBILITY:
Eligibility Criteria

1. Participants with differentiated thyroid cancer, non-RET-mutated medullary thyroid cancer, or poorly differentiated thyroid cancer who present with locoregionally advanced disease, as defined by extrathyroidal and/or extra nodal extension, or with advanced recurrent/residual invasive/bulky nodal disease will be enrolled in this trial, regardless of whether distant metastases are present or not.
2. At least 18 years of age on the day of signing informed consent.
3. Pathologic findings supporting the clinical impression of papillary thyroid cancer, follicular thyroid cancer, oncocytic thyroid cancer, medullary thyroid carcinoma, and/or poorly differentiated thyroid carcinoma.
4. Surgical morbidity/complexity score of 1 to 4 (moderate, severe, very severe, or unresectable).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 with no known sudden deterioration 2 weeks prior to the first dose of trial treatment.
6. Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs), including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (e.g., physiological replacement of mineral corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy are permitted.
7. Adequate organ and marrow function, based upon meeting all the following laboratory criteria within 28 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC)≥ 1500/mm3 (≥1.5 GI/L) without granulocyte colony-stimulating factor support within 2 weeks of screening laboratory sample collection.
   2. Platelets ≥ 100,000/mm3 (≥100 GI/L) without transfusion within 2 weeks of screening laboratory sample collection.
   3. Hemoglobin ≥9 g/dL (≥90 g/L) without transfusion within 2 weeks prior to screening laboratory sample collection.
   4. International Normalized Ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.2 x upper limit of normal (ULN).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x ULN. For subjects with documented bone metastasis ALP ≤5 x ULN.
   6. Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert fs disease ≤ 3 x ULN).
   7. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40 mL/min ( ≥0.67 mL/sec) using the Cockcroft Gault equation.
   8. Urine protein-to-creatinine ratio (UPCR) ≤1 mg/mg ( ≤113.2 mg/mmol) creatinine.
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
9. For MD Anderson site only, subjects must be willing to undergo tumor biopsy prior to trial treatment, unless in the opinion of the treating physician, a biopsy is not feasible or safe. For all sites, subjects must be willing to ultimately undergo surgery if their tumor becomes surgically resectable. Subjects retain the right to refuse any research interventions.
10. Sexually active fertile subjects and their partners must agree to use highly effective method of contraception (defined in Appendix A) during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (e.g., condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods. (1) through 186 days after the last dose of zanzalintinib for women of childbearing potential (WOCBP) or through 96 days after the last dose of zanzalintinib for men.
11. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.

Exclusion Criteria:

1. Medullary thyroid cancer participants with germline RET or known somatic RET mutations.
2. Prior treatment with zanzalintinib.
3. Prior treatment with a tyrosine kinase inhibitor.
4. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
5. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
7. Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin inhibitors) and platelet inhibitors (e.g., clopidogrel).

   Allowed anticoagulants are the following:
   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.

   Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
8. Any complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
9. The participant has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Unstable or deteriorating cardiovascular disorders: i. Congestive heart failure New York Heart Association class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g., ventricular flutter, ventricular fibrillation, Torsades de pointes). ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.

   iv. Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before to first dose of study treatment. Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Participants who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.
10. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
11. Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed. Intratracheal disease is allowed, as long as the endotracheal disease is not associated with major bleeding episodes.
12. Lesions invading major blood vessel including, but are not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Subjects with internal jugular vein involvement or tumor thrombus in the neck are eligible. Additionally, subjects with intravascular tumor extension (e.g., tumor thrombus in renal vein or inferior V. cava) may be eligiblefollowing Principal Investigator approval.
13. Other clinically significant disorders that would preclude safe study participation.

    1. Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.
    2. Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)- related illness except for subjects meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) CD4+ T cell count ≥ 200/μL; and (3) an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: To be eligible, participants taking CYP inhibitors (e.g., zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts and viral load are monitored per standard of care by the local health care provider.
    3. Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
    4. Malabsorption syndrome.
    5. Uncontrolled symptomatic hyperthyroidism or hypothyroidism.
    6. Uncontrolled symptomatic hypercalcemia or hypocalcemia.
    7. Moderate to severe hepatic impairment (Child-Pugh B or C).
    8. Requirement for hemodialysis or peritoneal dialysis.
    9. History of solid organ or allogeneic stem cell transplant.
14. Major surgery (as defined in Appendix B; e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Minor surgery (e.g., simple excision, tooth extraction) within 5 days before first dose of study treatment. Fine needle aspiration and core biopsies are allowed on study drug without drug hold.Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

    Note: Participants with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
15. Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment.

    Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
16. History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
17. Pregnant or lactating females.
18. Inability to swallow tablets or ingest a suspension either orally or by nasogastric (NG) or gastrostomy (PEG) tube.
19. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
20. Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to Investigational Product, within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
21. Other conditions, which in the opinion of the Investigator, would compromise the safety of the participant or the participants ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zafereo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org